CLINICAL TRIAL: NCT00045682
Title: A Phase II Evaluation of CT-2103 in the Third-Line Treatment of Recurrent or Persistent Epithelial Ovarian or Primary Peritoneal Cancer
Brief Title: CT-2103 in Treating Patients With Recurrent or Persistent Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0186C; NCI-2012-02493 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000257039; GOG-0186C (Other: Gynecologic Oncology Group); GOG-0186C (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Primary Peritoneal Carcinoma; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — paclitaxel poliglumex

ARMS (1):
- Treatment (polyglutamate paclitaxel) (Experimental): Patients receive polyglutamate paclitaxel (CT-2103) IV over 10-20 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel Poliglumex

INTERVENTIONS:
Drug: Paclitaxel Poliglumex — Given IV
  Other Names: CT-2103; Paclitaxel Polyglutamate; PG-TXL; Xyotax

SUMMARY:
Phase II trial to study the effectiveness of CT-2103 in treating patients who have recurrent or persistent ovarian epithelial cancer or primary peritoneal cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of polyglutamate paclitaxel (CT-2103) as third-line treatment for patients with recurrent or persistent ovarian epithelial or primary peritoneal cancer.

II. Determine the nature and degree of toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive polyglutamate paclitaxel (CT-2103) IV over 10-20 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or persistent ovarian epithelial cancer or primary peritoneal cancer after second-line therapy

  * Received 1 prior platinum-based first-line chemotherapy regimen and 1 prior second-line (non-platinum, non-taxane) chemotherapy regimen
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * At least 1 target lesion that has not previously been irradiated
* Ineligible for a higher priority GOG protocol (if one exists)
* Ineligible for the currently active phase II cytotoxic protocol for platinum-resistant disease
* Performance status - GOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No active bleeding
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* PT or PTT less than ULN
* Creatinine no greater than 1.5 times ULN
* No uncontrolled hypertension
* No uncompensated congestive heart failure
* No symptomatic coronary artery disease
* No myocardial infarction within the past 6 months
* No sensory or motor neuropathy greater than grade 1
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 3 weeks since prior biological therapy or immunotherapy directed at the malignancy
* No prior polyglutamate paclitaxel (CT-2103)
* Recovered from prior chemotherapy
* At least 1 week since prior hormonal therapy directed at the malignancy
* Concurrent hormone replacement therapy allowed
* Recovered from prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* Recovered from prior surgery
* At least 3 weeks since other prior therapy directed at the malignancy
* No prior therapy for another malignancy that would preclude this study
* No concurrent amifostine or other protective reagents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2002-09; Primary Completion 2006-07-15 (Actual)

PRIMARY OUTCOMES:
Frequency and duration of objective response | 5 years
Frequency and severity of observed adverse effects | 5 years
Survival time | 5 years
Duration of progression-free interval | 5 years

SECONDARY OUTCOMES:
Change in objective response | Baseline to 5 years
Change in observed adverse effects | Baseline to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States